CLINICAL TRIAL: NCT06882460
Title: Lifestyle Solutions to Postprandial Hypotension in Spinal Cord Injury
Brief Title: Diet and Exercise Solutions to Postprandial Hypotension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Ceren Yarar-Fisher, Principal Investigator, The Craig H. Neilsen Foundation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2024H0147
Record Dates: First submitted 2024-12-12; First posted 2025-03-18 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries
Keywords: postprandial hypotension; electrical stimulation; low-glycemic diet
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High glycemic load (Placebo Comparator)
  Interventions: Other: High glycemic load diet
- Low glycemic load (Experimental)
  Interventions: Other: Low glycemic load
- Electrical Stimulation (Experimental)
  Interventions: Other: Electrical stimulation exercise; Other: High glycemic load diet

INTERVENTIONS:
Other: Low glycemic load — Low glycemic load diet
  Arms: Low glycemic load
Other: Electrical stimulation exercise — Lower-body electrical stimulation exercise for 1-h after eating
  Arms: Electrical Stimulation
Other: High glycemic load diet — High glycemic load diet
  Arms: Electrical Stimulation; High glycemic load

SUMMARY:
The purpose of this study is to determine if a low glycemic diet and lower-body electrical stimulation can reduce postprandial hypotension in individuals with chronic spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury (SCI) between C4 and T12 who require use of wheelchair for daily mobility
* AIS A or B
* >1-year post-injury

Exclusion Criteria:

* Currently pregnant of breast-feeding
* Type 1 or 2 diabetes
* Previous gut augmentation bariatric surgery
* Neurological impairment other than SCI
* History of uncontrolled autonomic dysreflexia
* History of bone fractures
* Use of abdominal binder or anti-hypotensive drugs
* Fitted with pacemaker or defibrillator
* Currently receiving electrical stimulation training or in the previous year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Magnitude of systolic blood pressure decrease (in-lab) | Visit 2-4, Day 1
  Calculated as the maximum decrease in systolic blood pressure in the 2-h after eating breakfast and lunch under laboratory-controlled conditions

SECONDARY OUTCOMES:
Magnitude of systolic blood pressure decrease (at-home) | Visits 2-4, Days 1-3
  Calculated as the maximum decrease in systolic blood pressure in the 2-h after eating breakfast, lunch, and dinner for 3-days during at-home testing
Postprandial glucose (in-lab) | Visits 2-4, Day 1
  Blood samples will be obtained from an intravenous catheter at regular intervals after eating breakfast (3-h) and lunch (2-h) under laboratory controlled conditions.
Postprandial insulin (in-lab) | Visits 2-4, Day 1
  Blood samples will be obtained from an intravenous catheter at regular intervals after eating breakfast (3-h) and lunch (2-h) under laboratory controlled conditions.
Postprandial glucose (at-home) | Visits 2-4, Day 1-3
  A continuous glucose monitor will be used to measure glucose for 2-h after breakfast, lunch, and dinner for 3-days during at-home testing
Blood flow (in-lab) | Visits 2-4, Day 1
  Blood flow at the radial, brachial, popliteal and superior mesenteric arteries will be obtained using Doppler imaging at regular intervals after eating breakfast (3-h) and lunch (2-h) under laboratory controlled conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Dodd Rehabilitation Hospital, Columbus, Ohio, United States